CLINICAL TRIAL: NCT02854007
Title: REgistry of PAtients Treated With bioabsoRbable Devices in dAily Clinical Practice: Costs, Effectiveness, QALYs, and Efficiency. REPARA-QALY Registry
Brief Title: Costs, Effectiveness, QALYs, and Efficiency of Bioabsorbable Devices in Daily Clinical Practice
Acronym: REPARA-QALY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sección Hemodinamica y Cardiologia Intervencionista (Other)
Responsible Party: Sponsor
Other Study IDs: COR-BVS-2016-01
Record Dates: First submitted 2016-07-21; First posted 2016-08-03 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-07

CONDITIONS: Coronary Stenosis Treated With Implant of Bioresorbable Devices
Keywords: Coronary artery disease; Angioplasty; Bioresorbable coronary device; QALY (Quality-Adjusted Life Years)
MeSH Terms: conditions — Coronary Artery Disease | interventions — Angioplasty, Balloon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Coronary stenosis treated with Absorb: Patients with ischemic heart disease who have undergone percutaneous coronary revascularization with Absorb according to standard clinical practice. One thousand revascularized patients will be recruited at 40 siteS.
  Interventions: Device: Coronary angioplasty with implant of bioresorbable device

INTERVENTIONS:
Device: Coronary angioplasty with implant of bioresorbable device — Percutaneous coronary intervention

SUMMARY:
A multicenter, prospective, observational cohort study with clinical, quality of life, and economic evaluation to ascertain the quality-adjusted life years (QALYs) gained by patients with ischemic heart disease revascularized with Absorb in standard clinical practice in Spain. A before-after comparative analysis will be performed, so that each patient will act as his/her own control.

DETAILED DESCRIPTION:
Economical evaluation study of the efficiency of Absorb in a cohort of patients with ischemic heart disease who have undergone revascularization with Absorb based on the criteria established according to standard clinical practice. A comparison group without Absorb cannot be used for ethical reasons. Thus, each patient will act as his/her own control, and a before-after comparison will be done. This is therefore a prospective, observational cohort study with concurrent data collection.

Primary objective:

* To assess utility (QALYs gained) in patients implanted Absorb in standard clinical practice conditions.

Secondary objectives:

* To assess effectiveness (clinical outcomes) in patients who undergo coronary revascularization with Absorb implantation.
* To assess costs (direct and indirect) derived from coronary revascularization with Absorb implantation.
* To assess efficiency in terms of cost/utility (cost per QALY gained) and cost/effectiveness (cost per MACE -major cardiac adverse events- free patient).

ELIGIBILITY:
Inclusion Criteria:

* Age ranging from 18 and 95 years.
* Both sexes.
* Coronary revascularization with Absorb for any of the following lesions: de novo, restenosis, segment ST elevation myocardial infarction (STEMI), chronic total occlusion (CTO), trunk, venous graft, or bifurcations.
* Informed consent signed before participation in the study is started.

Exclusion Criteria:

* Pregnant or nursing woman..
* Cardiogenic shock.
* Refusal to participate in the study.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic heart disease who have undergone percutaneous coronary revascularization with Absorb according to standard clinical practice. One thousand revascularized patients will be recruited at 40 sites.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Quality Adjusted Live Years (QALYs) gained since the first revascularization (the week before revascularization) to the end of follow-up (one year) | 1 year follow-up
  To construct QALYs, the EuroQoL-5D-3L (EQ-5D) will be used for the quality of life dimension, while the time elapsed between each EQ-5D measurement will be considered for the time dimension. If a patient dies, the value of EQ-5D is 0 from the date of death.

SECONDARY OUTCOMES:
"Target lesion failure", defined as cardiac death, target-vessel myocardial infarction, and target lesion ischemia at any time during the follow-up period. | 1 year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Hernandez, MD, Principal Investigator — Hospital 12 de Octubre, Madrid
Locations (1):
- Hospital 12 de Octubre, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No